CLINICAL TRIAL: NCT06241196
Title: Vestibular Socket Therapy Using Acellular Dermal Matrix Versus Connective Tissue Graft in Immediate Implants of Aesthetic Zone
Brief Title: Vestibular Socket Therapy Using Acellular Dermal Matrix Versus Connective Tissue Graft
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Amr Anwar Mohamed Ellithy Yousef, Assistant lecturer, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Implant_22
Record Dates: First submitted 2023-06-19; First posted 2024-02-05 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-01

CONDITIONS: Immediate Implant
Keywords: vestibular socket therapy; dental implant; soft tissue graft
MeSH Terms: interventions — Mutagenesis, Insertional; Alloderm

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Group I (Active Comparator): Ten sites will be treated by immediate implant and VST with Alloderm + allogenic bone membrane and xenograft.
  Interventions: Device: implant; Procedure: Vestibular Socket Therapy; Drug: Alloderm; Drug: Xenogenic bone membrane shield
- Group II (Experimental): Ten sites will be treated by immediate implant and VST with connective tissue graft + allogenic bone membrane and xenograft.
  Interventions: Device: implant; Procedure: Vestibular Socket Therapy; Drug: Xenogenic bone membrane shield; Procedure: Connective tissue graft

INTERVENTIONS:
Device: implant — Implant will be placed through the surgical guide in the extraction socket
  Other Names: biohorizons implant, the pro,platform switching design,USA
Procedure: Vestibular Socket Therapy — tunnel incision will be made in labial vestibule
  Other Names: VST
Drug: Alloderm — allogenic soft tissue substitute
  Other Names: AlloDerm SELECT™ RTM,biohorizons
  Arms: Group I
Drug: Xenogenic bone membrane shield — xenogenic bone membrane
  Other Names: Osteobiol ,flexible xenograft cortical sheet from Technoss,USA
Procedure: Connective tissue graft — soft tissue harvesting from palate
  Other Names: CTG
  Arms: Group II

SUMMARY:
The aim of this study is to evaluate and compare the Vestibular Socket Therapy (VST) technique using alloderm versus connective tissue graft both with xenogenic bone membrane in immediate implants of anterior aesthetic zone.

DETAILED DESCRIPTION:
Twenty surgical sites will be divided into two groups; each of which has 10 surgical sites. Grouping will be done randomly sequentially numbered, opaque, sealed envelopes (SNOSE)

The groups will be treated as follow:

* Group I: Ten sites will be treated by immediate implant and VST with Alloderm + allogenic bone membrane and xenograft.
* Group II: Ten sites will be treated by immediate implant and VST with connective tissue graft + allogenic bone membrane and xenograft Each group will be subjected to intraoral scanning at baseline, 6 months and 12 months. The changes in peri-implant mucosal level will be assessed by superimposition of scanning files of different intervals to monitor the changes in surface area calculated by software.

The changes in gingival phenotype could be assessed at 6 months and 12 months intervals by superimposition of DICOM files on CBCT software Each group will be subjected to Cone Beam Computed Tomography (CBCT) at baseline, 6 months and 12months to asses both thickness and height of labial (facial) plate of bone and implant survival.

ELIGIBILITY:
Inclusion Criteria:

* Adults (20-50) years old.
* Class II socket according to Elian et al, (7)described as facial soft tissue is present but the buccal plate is partially missing following extraction of the tooth in the maxillary anterior region.
* Thin gingival phenotype.
* Bone quality ranges from D2-D3 as gained from preoperative cone beam computed tomography.
* Presence of at least 3 mm of keratinized gingiva.
* Optimal compliance as evidenced by no missing treatment appointments and positive attitude towards oral hygiene.

Exclusion Criteria:

* Medically compromised patients and systemic conditions precluding implant and periodontal surgery.
* Smokers, diabetics, pregnant or lactating women.
* History of chemotherapy, radiotherapy in head and/or neck region.
* Bisphosphonate therapy.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
changes in peri-implant mucosal level | baseline, 6, 12 months
  level of peri-implant mucosa
changes in gingival phenotype | baseline, 6, 12 months
  thickness of peri-implant mucosa

SECONDARY OUTCOMES:
thickness of labial (facial) plate of bone | baseline, 6, 12 months
  three area measures of facial bone
implant survival | baseline, 6, 12 months
  implant stability, health, mobility and function
height of labial (facial) plate of bone | baseline, 6, 12 months
  Apico-coronal height of labial bone

CONTACTS AND LOCATIONS:
Overall Officials: amr anwar mohammed ellithy yousef, Msc, Principal Investigator — Tanta University
Locations (1):
- TantaU, Tanta, Gharbia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol (2022-04-10): https://cdn.clinicaltrials.gov/large-docs/96/NCT06241196/Prot_000.pdf